CLINICAL TRIAL: NCT07016451
Title: Low-intensity Extracorporeal Shockwaves in the Treatment of Radiation Cystitis, Randomized Controlled Trial
Brief Title: Efficacy of Low-Intensity Shockwave Therapy in Treating Radiation Cystitis
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Thanakrit Visuthikosol (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor-Investigator, Thanakrit Visuthikosol, Thanakrit Visuthikosol, MD, Ramathibodi Hospital
Organization: Ramathibodi Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MURA2023/837
Record Dates: First submitted 2025-05-13; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Radiation Cystitis
Keywords: Radiation cystitis; Li-ESWT
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patient receives the treatment, medication or intervention that not included Li-ESWT
  Interventions: Drug: Medication
- Li-ESWT (Experimental): The intervention treatment for Radiation cystitis mainly or only uses Li-ESWT. If the patients have regular medication for this disease, they will receive continuous treatment
  Interventions: Procedure: Li-ESWT; Drug: Medication

INTERVENTIONS:
Procedure: Li-ESWT — The intervention treatment uses Li-ESWT. (Dornier Aries® devices, Power 0.29mj/m² and 3000 shocks per week for 4 weeks)
  Arms: Li-ESWT
Drug: Medication — The medication treatment of Radiation cystitis and relevant symptoms such as Antimuscarinics, Beta3 agonist, and pain control, as listed. Antimuscarinic Agents
  * Oxybutynin
  * Tolterodine
  * Solifenacin
  * Darifenacin
  * Trospium
  * Fesoterodine β3-Adrenergic Agonists
  * Mirabegron Pain Control Medications
  * Paracetamol
  * NSAIDs (e.g., Ibuprofen, Diclofenac)
  * Phenazopyridine
  * Amitriptyline
  * Gabapentin / Pregabalin

SUMMARY:
Radiation-induced cystitis is a condition commonly seen in patients who have undergone radiation therapy, especially those treated in the pelvic region. Symptoms typically manifest after radiation exposure and may include dysuria (painful urination), increased urinary frequency during both day and night, and hematuria (blood in the urine), which can range from mild to severe.

Currently, treatment is symptomatic, as there is no definitive cure for radiation cystitis. Management includes medications to alleviate symptoms, cystoscopic interventions to control bleeding, intravesical instillations, and in severe cases, surgical procedures to divert the urinary tract.

Recently, low-intensity extracorporeal shock wave therapy (Li-ESWT) has been used to treat various urological conditions, including chronic prostatitis, chronic cystitis, overactive bladder, erectile dysfunction, and as an adjunct to enhance drug delivery into the bladder. This modality has shown potential to reduce inflammation, promote angiogenesis (formation of new blood vessels), regenerate tissues, and restore neural function.

For patients with radiation cystitis, particularly those with prostate cancer who have received pelvic radiation, shock wave therapy is being explored for its ability to alleviate bladder pain and inflammation. This approach is similar to its use in non-bacterial cystitis and overactive bladder conditions.

Studies have identified elevated levels of specific proteins in the urine of patients with radiation-induced cystitis, including markers of fibrosis, angiogenesis, and inflammation, which differ from those found in non-irradiated individuals.

The anticipated benefit of this study is to provide data on clinical symptoms and treatment safety, potentially offering a novel therapeutic strategy for managing radiation-induced cystitis.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for diagnosis of radiation-induced cystitis and a history of pelvic radiation therapy administered more than 6 months prior.
* Aged 18 years or older.
* Willing to participate in the research study by providing written informed consent.

Exclusion Criteria:

* Active urinary tract infection within the past 6 months.
* Active and uncontrolled gross hematuria.
* Patients currently have a urinary diversion or abdominal ostomy.
* Patients with anuria due to chronic kidney failure.
* Uncontrolled coagulopathy.
* Refuse participation, withdraw from the study, or experience severe adverse effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms | Before, 1, and 3 months after treatment
  In each study group, comparative analysis of symptoms such as urination frequency, nocturia, dysuria, and incontinence is conducted before and after treatment.
  Each parameter is recorded by the patient in a bladder diary, capturing the frequency and intensity of symptoms experienced daily for the preceding three days.

SECONDARY OUTCOMES:
Urine Molecular Analysis | Before, 1, and 3 months after treatment
  Report the number and compare before and after treatment. Each study patient group's molecular analysis of inflammation, fibrosis, and vasculogenesis.
  Fibrosis: PAI 1, TIMP1, and TIMP2 inflammatory: IL-1a, IL-6, and MIP-1a Vascular maker: HGF, and VEGF-A

OTHER OUTCOMES:
Urine analysis | Before, 1, and 3 months after treatment
  Urine analysis for WBC, RBC, and protein

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
We are still evaluating whether to share individual participant data (IPD) from this study on low-intensity extracorporeal shock wave therapy (Li-ESWT) for radiation-induced cystitis. Key considerations include ensuring adequate de-identification of sensitive clinical data, addressing patient consent for secondary use, and complying with institutional and ethical guidelines. Additionally, due to the relatively small sample size and the potential for indirect re-identification, we are carefully assessing the risks and benefits of IPD sharing. A decision will be made once these factors have been thoroughly reviewed in consultation with our ethics board and institutional data governance policies.